CLINICAL TRIAL: NCT03428126
Title: Phase II Study of Durvalumab (MEDI4736) (Anti-PD-L1) and Trametinib (MEKi) in MSS Metastatic Colon Cancer
Brief Title: Study of Durvalumab (MEDI4736) (Anti-PD-L1) and Trametinib (MEKi) in MSS Metastatic Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0514; NCI-2018-00911 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Malignant Neoplasms of Digestive Organs; Colorectal Cancer; Colon Cancer
Keywords: Malignant neoplasms of digestive organs; Colorectal Cancer; Colon Cancer; Durvalumab; MEDI4736; Trametinib; GSK1120212
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — durvalumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Trametinib (Experimental): Participants take Trametinib tablets by mouth every day. Trametinib taken alone for the first 7 days of the study then participants begin receiving it in combination with Durvalumab.
  Participants receive Durvalumab by vein every 4 weeks.
  Each cycle is 28 days.
  Interventions: Drug: Durvalumab; Drug: Trametinib

INTERVENTIONS:
Drug: Durvalumab — Dose Escalation and Dose Expansion Dose: 1500 mg by vein every 4 weeks in a 28 day cycle.
  Other Names: MEDI4736
Drug: Trametinib — Dose Escalation Starting Dose: 2mg by mouth daily in a 28 day cycle.
  Dose Expansion Dose: MTD from Dose Escalation.
  Other Names: GSK1120212

SUMMARY:
The goal of this clinical research study is to learn if durvalumab and trametinib can help to control microsatellite stable (MSS) colorectal cancer. The safety of these drugs will also be studied.

This is an investigational study. Durvalumab is FDA approved and commercially available for the treatment of previously treated advanced bladder cancer. Trametinib is FDA approved in combination with another drug called dabrafenib for the treatment of unresectable or metastatic melanoma with BRAF V600E or BRAF V600K.

It is investigational to use durvalumab and trametinib to treat MSS colorectal cancer.

Up to 56 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle is 28 days.

Participant will take trametinib tablets by mouth every day with at least 8 ounces of water. Each dose should be taken at about the same time each day, 1 hour before or 2 hours after a meal. Participant should not crush, cut, or chew the tablets. If participant misses a dose of trametinib, participant may take the tablets as soon as participant remembers but only if participant's next scheduled dose is at least 12 hours later. If participant's next scheduled dose is less than 12 hours, participant should wait and take participant's next dose as scheduled.

Participant will take trametinib alone for the first 7 days of the study and then participant will begin receiving it in combination with durvalumab.

Every 4 weeks, participant will receive durvalumab by vein over about 60 minutes.

Length of Treatment:

Participant will be able to receive the study drugs for as long as the doctor thinks it is in participant's best interest. Participant no longer will take the study drugs if intolerable side effects occur or if the study doctor decides that the drugs are no longer working.

It is expected that participation in this study may last about 12 months.

Participation in this study will be over after follow-up.

Study Visits:

On Day 1 of Weeks 0, 2, 4, 6, 12, and then every 4 weeks after that (Weeks 16, 20, 24, and so on):

* Participant will have a physical exam.
* Blood (about 6 tablespoons) will be drawn for routine tests, immune system testing, and biomarker testing.
* If participant had a biopsy at screening, participant will have another biopsy during Week 4 to check the status of the disease and for biomarker testing. Depending on when participant joins the study, this biopsy may be optional.

On Day 1 of Week 8:

* Participant will have a physical exam.
* Blood (about 6 tablespoons) will be drawn for routine tests, immune system testing, and biomarker testing.
* Participant will have a CT scan.

On Day 1 of Week 16 and then every 8 weeks after that (Weeks 24, 32, 40, and so on), participant will have a CT scan.

End-of-Treatment:

About 28 days after participant's last dose of study drugs, participant will have a physical exam.

Follow-Up:

After participant's end-of-treatment visit, participant will be called by the study staff every 3 months for up to 18 months to ask how participant is doing. Each call should last about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed metastatic colorectal cancer.
2. Patients must have measurable disease per RECIST v1.1 criteria.
3. Patients must have had at least prior treatment with a fluoropyrimidine and either oxaliplatin or irinotecan.
4. Age >/=18 years. Because no dosing or adverse event data are currently available on the use of this combination in patients <18 years of age, children are excluded from this study.
5. Body weight > 30kg.
6. Life expectancy of greater than 6 months.
7. ECOG performance status 0-1 (Karnofsky >/=70%).
8. Patients must have normal organ and marrow function as defined below: - Leukocytes >/=3,000/mcL, Absolute neutrophil count >/=1,500/mcL, Hemoglobin >/=9.0g/dL, Platelets >/=75,000/mcL, Total bilirubin < 1.5 X institutional normal limits (subjects with known Gilbert syndrome are eligible with total bilirubin < 3.0 mg/dL), AST(SGOT)/ALT(SGPT) </=2.5 X institutional ULN (</= 5 if liver metastases present), Creatinine within normal institutional limits OR, Creatinine clearance > 40mL/min by Cockcroft-Gault or 24h urine collection.
9. Known MSS status by either IHC or PCR. Known or evaluable BRAF and KRAS status.
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: -- Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
11. Inclusion #10 cont'd -- Women >/=50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
12. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately and will be removed from the study.
13. Ability to understand and the willingness to sign a written informed consent document.
14. Willingness to have 2 tumor biopsies; the first before and the second while on therapy (optional for all patients and may become mandatory in order to ensure 15 patients at MTD have paired biopsies).

Exclusion Criteria:

1. Patients who have had chemotherapy within 2 weeks prior to first dose of study drug.
2. Any unresolved toxicity NCI CTCAE Grade >/=2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria: -- Subjects with Grade >/=2 neuropathy will be evaluated on a case-by-case basis after consultation with the Principal investigator.-- Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Principal investigator.
3. Patients may not be receiving any other investigational agents.
4. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medication. Note: Local surgery of isolated lesions for palliative intent is acceptable.
5. Patients with known brain metastases or leptomeningeal carcinomatosis will be excluded from this clinical trial. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
6. Mean QT interval corrected for heart rate (QTc) >/= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
7. History of pneumonitis or interstitial lung disease (ILD).
8. History of allogenic organ transplantation.
9. Subjects with active, known, or suspected autoimmune disease including patients with a history of inflammatory bowel disease (ulcerative colitis or Crohn's disease); patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis), and central nervous system or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome, myasthenia gravis, multiple sclerosis). Subjects with vitiligo, type I diabetes mellitus, Grave's disease, Hashimoto thyroiditis, psoriasis, and other mild autoimmune disease not requiring systemic treatment are permitted to enroll at the discretion of the investigator.
10. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
11. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
12. Prior exposure to T cell checkpoint inhibitor therapies.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. History of active primary immunodeficiency.
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice for patients suspected of having active infection), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of study medications.
17. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Johnson B, Haymaker CL, Parra ER, Soto LMS, Wang X, Thomas JV, Dasari A, Morris VK, Raghav K, Vilar E, Kee BK, Eng C, Parseghian CM, Wolff RA, Lee Y, Lorenzini D, Laberiano-Fernandez C, Verma A, Lang W, Wistuba II, Futreal A, Kopetz S, Overman MJ. Phase II study of durvalumab (anti-PD-L1) and trametinib (MEKi) in microsatellite stable (MSS) metastatic colorectal cancer (mCRC). J Immunother Cancer. 2022 Aug;10(8):e005332. doi: 10.1136/jitc-2022-005332. PMID 36007963
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 patients were enrolled to the first stage at The University of Texas MD Anderson Cancer Center.
Groups:
- Durvalumab + Trametinib: Single arm study. All participants received both study drugs
Period: Overall Study
Arm/Group | Durvalumab + Trametinib
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab + Trametinib
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 48 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Single arm study. All study participants received both study drugs.
  Participants
    Female | 14
    Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Single arm study. All study participants received both study drugs.
  Participants
    Hispanic or Latino | 3
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants] — Single arm study. All study participants received both study drugs.
  Participants
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 21
    More than one race | 0
    Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants] — Single arm study. All study participants received both study drugs.
  participants
    United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Best Overall Response Rate.
Description: Best overall response rate (CR+PR) by immune-related response rate.
Time Frame: From Baseline to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab + Trametinib: Single arm study. All study participants received both study drugs.
Arm/Group | Durvalumab + Trametinib
Number analyzed (Participants) | 29
Participants | 1

2. Secondary Outcome: Progression Free Survival as Determined by irRC
Description: The Kaplan-Meier method GraphPad software, V.8 was used for statistical analyses.
Time Frame: From Baseline to up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + Trametinib
Number analyzed (Participants) | 29
months | 3.2 [2.5 to 3.8]

3. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method GraphPad software, V.8 was used for statistical analyses.
Time Frame: From Baseline to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Durvalumab + Trametinib: Singe arm study. All participants received both study drugs.
Arm/Group | Durvalumab + Trametinib
Number analyzed (Participants) | 29
months | 6.9 [5.7 to 8]

4. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) describes the percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response, partial response, or stable disease.
Time Frame: From Baseline to 2 years.
Measure: Number; unit: percentage
Arm/Group | Durvalumab + Trametinib
Number analyzed (Participants) | 29
percentage
  Complete Response | 0
  Partial Response | 3.4
  Stable Disease | 24

ADVERSE EVENTS:
Time Frame: from Baseline to 2 years
Arm/Group | Durvalumab + Trametinib
All-Cause Mortality (participants affected / at risk) | 12/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab + Trametinib (N=29)
Fatigue (General disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 25
Anorexia (Gastrointestinal disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Alanine aminotransferase (Investigations) | 7
Bilirubin (Investigations) | 2
Aspartrate aminotransferase (Investigations) | 9
Alkaline phosphatase (Investigations) | 11
Anemia (Investigations) | 12
Thrombocytopenia (Investigations) | 8
Lipase (Investigations) | 6
Amylase (Investigations) | 5
Hypothyroidism (Investigations) | 3
Hyponatremia (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03428126/Prot_SAP_000.pdf